CLINICAL TRIAL: NCT04181827
Title: A Phase 3 Randomized Study Comparing JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA, Versus Pomalidomide, Bortezomib and Dexamethasone (PVd) or Daratumumab, Pomalidomide and Dexamethasone (DPd) in Subjects With Relapsed and Lenalidomide-Refractory Multiple Myeloma
Brief Title: A Study Comparing JNJ-68284528, a CAR-T Therapy Directed Against B-cell Maturation Antigen (BCMA), Versus Pomalidomide, Bortezomib and Dexamethasone (PVd) or Daratumumab, Pomalidomide and Dexamethasone (DPd) in Participants With Relapsed and Lenalidomide-Refractory Multiple Myeloma
Acronym: CARTITUDE-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108695; 68284528MMY3002 (Other: Janssen Research & Development, LLC); 2019-001413-16 (EudraCT Number); 2023-506588-32-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: PVd or DPd (Standard Therapy) (Experimental): Participants will receive either PVd or DPd as a standard therapy. In PVd treatment, participants will receive oral pomalidomide 4 mg on Days 1 to 14 in each cycle; bortezomib 1.3 mg/meter square (m^2) SC on Days 1, 4, 8 and 11 (Cycles 1 to 8) and on Days 1 and 8 (Cycle 9 onwards) and oral dexamethasone 20 mg on Days 1, 2, 4, 5, 8, 9, 11 and 12 (Cycles 1 to 8) and Days 1, 2, 8 and 9 (Cycle 9 onwards). Each cycle will consist of 21 days. In DPd treatment, participants will receive daratumumab SC 1800 mg weekly on Days 1, 8, 15, and 22 (Cycles 1 and 2), every 2 weeks on Days 1 and 15 (Cycles 3 to 6) and every 4 weeks on Day 1 (Cycle 7 onwards); oral pomalidomide 4 mg on Days 1 to 21 (Cycle 1 onwards); dexamethasone 40 mg oral or IV weekly on Days 1, 8, 15, and 22 (Cycle 1 onwards). Each cycle will consist of 28 days. Participants will continue to receive PVd or DPd until confirmed PD, death, intolerable toxicity, withdrawal of consent, or end of the study, whichever occurs earlier.
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Daratumumab
- Arm B: (Ciltacabtagene Autoleucel [Cilta-cel]) (Experimental): Participants will receive at least one cycle of bridging therapy (PVd or DPd) and additional cycles of bridging therapy may be considered based on participant's clinical status and timing of availability of cilta-cel along with conditioning regimen (cyclophosphamide 300 milligram [mg]/m^2 intravenous [IV] and fludarabine 30 mg/m^2 IV daily, for 3 days), and cilta-cel infusion 0.75 * 10^6 chimeric antigen receptor (CAR)-positive viable T cells/ kilogram (kg).
  Interventions: Drug: Cilta-cel

INTERVENTIONS:
Drug: Cilta-cel — Cilta-cel infusion will be administered at a target dose of 0.75 * 10^6 CAR-positive viable T cells/kilogram (kg).
  Arms: Arm B: (Ciltacabtagene Autoleucel [Cilta-cel])
Drug: Pomalidomide — Pomalidomide 4 mg will be administered orally.
  Arms: Arm A: PVd or DPd (Standard Therapy)
Drug: Bortezomib — Bortezomib 1.3 milligram per meter square (mg/m^2) will be administered subcutaneously (SC).
  Arms: Arm A: PVd or DPd (Standard Therapy)
Drug: Dexamethasone — Dexamethasone 20 mg/day (10mg/day for participants >75 years of age) (on bortezomib treatment days and the days following bortezomib treatment) will be administered orally in PVd treatment; and orally or intravenous (IV) at 40 mg weekly (20mg weekly for participants >75 years of age) in DPd treatment.
  Arms: Arm A: PVd or DPd (Standard Therapy)
Drug: Daratumumab — Daratumumab 1800 mg will be administered SC.
  Arms: Arm A: PVd or DPd (Standard Therapy)

SUMMARY:
The purpose of this study is to compare the efficacy of ciltacabtagene autoleucel (cilta-cel) with standard therapy, either Pomalidomide, Bortezomib and Dexamethasone (PVd) or Daratumumab, Pomalidomide and Dexamethasone (DPd).

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease at screening as defined by any of the following: (a) Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 0.5 gram per deciliter (g/dL) or urine M-protein level >=200 milligram (mg)/24 hours; or (b) Light chain multiple myeloma without measurable M-protein in the serum or the urine: Serum free light chain >=10 mg/dL and abnormal serum free light chain ratio
* Have received 1 to 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD)
* Have documented evidence of PD by International Myeloma Working Group (IMWG) criteria based on investigator's determination on or within 6 months of their last regimen
* Be refractory to lenalidomide per IMWG consensus guidelines (failure to achieve minimal response or progression on or within 60 days of completing lenalidomide therapy). Progression on or within 60 days of the last dose of lenalidomide given as maintenance will meet this criterion. For participants with more than 1 prior line of therapy, there is no requirement to be lenalidomide refractory to the most recent line of prior therapy. However, participants must be refractory to lenalidomide in at least one prior line
* Have clinical laboratory values meeting the following criteria during the Screening Phase (re testing is allowed but the below criteria must be met in the latest test prior to randomization):

  1. Hemoglobin >=8 gram per deciliter (g/dL) (without prior RBC transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted);
  2. Absolute neutrophil count (ANC) >=1 * 10^9 per liter (L) (without recombinant human granulocyte colony-stimulating factor [G-CSF] within 7 days and without pegylated G-CSF within 14 days of the laboratory test);
  3. Platelet count >=75 * 10^9/L (without prior platelet transfusion within 7 days before the laboratory test) in participants in whom less than (<) 50 percent (%) of bone marrow nucleated cells are plasma cells; platelet count >=50 * 10^9/L (without prior platelet transfusion within 7 days before the laboratory test) in participants in whom >=50% of bone marrow nucleated cells are plasma cells;
  4. Lymphocyte count >=0.3 * 10^9/L;
  5. Aspartate aminotransferase (AST) less than or equal to (<=)3 * upper limit of normal (ULN);
  6. Alanine aminotransferase (ALT) <=3 * ULN;
  7. Total bilirubin <=2.0 * ULN; except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin <=1.5 * ULN is required);
  8. Estimated glomerular filtration rate >=40 milliliter per minute (mL/min) per 1.73 meter square (m^2) (to be calculated using the Modification of Diet in Renal Disease [MDRD] formula)

Exclusion Criteria:

* Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy directed at any target
* Any previous therapy that is targeted to B-cell maturation antigen (BCMA)
* Ongoing toxicity from previous anticancer therapy that has not resolved to baseline levels or to Grade 1 or less; except for alopecia
* Participants with Grade 1 peripheral neuropathy with pain or Grade 2 or higher peripheral neuropathy will not be permitted to receive pomalidomide, bortezomib, and dexamethasone (PVd) as standard therapy or bridging therapy; however, participants may receive daratumumab, pomalidomide, and dexamethasone (DPd) as standard therapy or bridging therapy
* Received a cumulative dose of corticosteroids equivalent to >=70 mg of prednisone within the 7 days prior to randomization
* Monoclonal antibody treatment within 21 days
* Cytotoxic therapy within 14 days
* Proteasome inhibitor therapy within 14 days
* Immunomodulatory drug (IMiD) therapy within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2029-04-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (88):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Cancer Center-Scottsdale, Phoenix, Arizona
  - Stanford University Medical Center, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - University Of Miami Leonard M Mille School Of Medicine SCCC, Miami, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Westwood, Kansas
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Wisconsin Institutes for Medical Research, Madison, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - Royal Brisbane and Womens Hospital, Herston
  - Peter MacCallum Cancer Centre, Melbourne
  - Alfred Health, Melbourne
  - Fiona Stanley Hospital, Murdoch
- Belgium (4):
  - Universitair Ziekenhuis - Antwerpen, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Rigshospitalet, Copenhagen, Denmark
- France (7):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - C.H.U. Hotel Dieu - France, Nantes
  - Hopital Saint Louis, Paris
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Germany (6):
  - Universitaetsklinikum Koeln, Cologne
  - Universitatsklinikum Carl Gustvav Carus Dresden an der Technischen Universitat Dresden, Dresden
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Eberhard Karls Universitaet Abt fur innere Med II Haematologie Onkologie Germany, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
- Attikon University General Hospital of Attica, Athens, Greece
- Israel (3):
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - IRCCS Ospedale San Raffaele HSR, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Policlinico Universitario Agostino Gemelli, Roma
  - A.O.U. Citta della Salute e della Scienza di Torino - Presidio Molinette, Turin
- Japan (8):
  - Kyushu University Hospital, Fukuoka
  - Kanazawa University Hospital, Kanazawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nagoya City University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya City
- Netherlands (4):
  - VU Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut BadawczyOddz w Gliwicach, Gliwice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Instytut Hematologii i Transfuzjologii, Warsaw
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (7):
  - Inst. Cat. D'Oncologia-Badalona, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Virgen Del Rocio, Seville
- Sweden (3):
  - Skane University Hospital, Lund
  - Karolinska Universitetssjukhuset Huddinge, Hematologiska Kliniken, Huddinge, Stockholm
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - University Hospital Wales, Cardiff
  - University College Hospital, London
  - Kings College Hospital, London
  - Christie Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Lopez-Munoz N, Bar N, Diels J, van Sanden S, Mendes J, Lee S, Hernando T, Lendvai N, Patel N, Ishida T, Er J, Harrison SJ. Ciltacabtagene Autoleucel Versus Idecabtagene Vicleucel in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma with 2-4 Prior Lines of Therapy: Updated Matching-Adjusted Indirect Comparison. Adv Ther. 2026 Feb 2. doi: 10.1007/s12325-025-03479-y. Online ahead of print. PMID 41627370
- [Derived] Einsele H, San-Miguel J, Dhakal B, Touzeau C, Leleu X, van de Donk NW, Sidana S, Oriol A, Cohen YC, Harrison SJ, Mateos MV, Martinez-Lopez J, Corradini P, Karlin L, Chen D, Li Q, Yeh TM, Li K, Plaks V, Slaughter A, Lonardi C, Benachour N, Ghosh A, Vogel M, Schecter JM, Lendvai N, Koneru M, Patel N, Florendo E, Ho PJ, Popat R. Cilta-cel in lenalidomide-refractory multiple myeloma (CARTITUDE-4): an updated analysis including overall survival from an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2026 Feb;27(2):254-268. doi: 10.1016/S1470-2045(25)00653-9. Epub 2026 Jan 7. PMID 41519141
- [Derived] Touzeau C, Lipe B, Khan AM, Dhakal B, Nair S, He J, Mendes J, Lee S, Lonardi C, Slaughter A, Lendvai N, Schecter JM, Chen D, Zhao M, Yeh TM, Leleu X, Puig N, Dytfeld D, Zamagni E, Weisel K, Karlin L, Delforge M, Corradini P, Mina R, Roeloffzen W, Sidana S. Comparative Effectiveness of Ciltacabtagene Autoleucel in CARTITUDE-4 Versus Real-World Physician's Choice of Therapy from the Flatiron Registry in Lenalidomide-Refractory Multiple Myeloma. Adv Ther. 2025 Oct;42(10):5023-5041. doi: 10.1007/s12325-025-03308-2. Epub 2025 Aug 6. PMID 40768190
- [Derived] Fonseca R, Diels J, Ghilotti F, Mendes J, Van Hoorenbeeck S, Lee S, Schecter JM, Lendvai N, Patel N, Triguero A, Alsdorf W, van de Donk NWCJ, Ursi M. Survival Outcomes with Cilta-cel Versus Conventional Treatment Regimens for Patients with Lenalidomide-Refractory Multiple Myeloma Using Inverse Probability of Treatment Weighting. Adv Ther. 2025 Sep;42(9):4418-4431. doi: 10.1007/s12325-025-03278-5. Epub 2025 Jul 4. PMID 40613875
- [Derived] Harrison SJ, Touzeau C, Kint N, Li K, Nguyen T, Mayeur-Rousse C, Rahman M, Le Bris Y, Er J, Eugene-Lamer J, Haynes NM, Li J, Abbott RC, Bodet-Milin C, Moreau A, Letouze E, Lendvai N, Schecter JM, Deraedt W, Banerjee A, Lengil T, Vogel M, Foulk B, Zhao H, Smirnov D, Slaughter A, Lonardi C, Lee E, Marquez L, Sankari A, Plaks V, Filho JOC, Patel N, Geng D, Gastinne T, Kelly H, Tiong IS, Eveillard M, Chevallier P, Lade S, Moreau P, Grimmond S, Oliaro J, Tessoulin B, Blombery P. CAR+ T-Cell Lymphoma after Cilta-cel Therapy for Relapsed or Refractory Myeloma. N Engl J Med. 2025 Feb 13;392(7):677-685. doi: 10.1056/NEJMoa2309728. PMID 39938094
- [Derived] Mina R, Mylin AK, Yokoyama H, Magen H, Alsdorf W, Minnema MC, Shune L, Isufi I, Harrison SJ, Shah UA, Schecter JM, Vogel M, Lendvai N, Gries KS, Katz EG, Slaughter A, Lonardi C, Gilbert J, Li Q, Deraedt W, Filho OC, Patel N, Florendo E, Karlin L, Weisel K. Patient-reported outcomes following ciltacabtagene autoleucel or standard of care in patients with lenalidomide-refractory multiple myeloma (CARTITUDE-4): results from a randomised, open-label, phase 3 trial. Lancet Haematol. 2025 Jan;12(1):e45-e56. doi: 10.1016/S2352-3026(24)00320-X. PMID 39756844
- [Derived] San-Miguel J, Dhakal B, Patel N, Schecter JM, Lendvai N, Einsele H. Plain language summary of the CARTITUDE-4 study of ciltacabtagene autoleucel for the treatment of people with relapsed or refractory multiple myeloma. Future Oncol. 2024;20(33):2509-2520. doi: 10.1080/14796694.2024.2376973. Epub 2024 Aug 7. PMID 39110421
- [Derived] San-Miguel J, Dhakal B, Yong K, Spencer A, Anguille S, Mateos MV, Fernandez de Larrea C, Martinez-Lopez J, Moreau P, Touzeau C, Leleu X, Avivi I, Cavo M, Ishida T, Kim SJ, Roeloffzen W, van de Donk NWCJ, Dytfeld D, Sidana S, Costa LJ, Oriol A, Popat R, Khan AM, Cohen YC, Ho PJ, Griffin J, Lendvai N, Lonardi C, Slaughter A, Schecter JM, Jackson CC, Connors K, Li K, Zudaire E, Chen D, Gilbert J, Yeh TM, Nagle S, Florendo E, Pacaud L, Patel N, Harrison SJ, Einsele H. Cilta-cel or Standard Care in Lenalidomide-Refractory Multiple Myeloma. N Engl J Med. 2023 Jul 27;389(4):335-347. doi: 10.1056/NEJMoa2303379. Epub 2023 Jun 5. PMID 37272512

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Currently results are reported until the primary completion date (01-May-2024). Results of remaining duration of the study will be reported after study completion.
Groups:
- Arm A: Standard Therapy: PVd or DPd: Participants received either PVd or DPd as standard therapy. In pomalidomide, bortezomib and dexamethasone (PVd) treatment, participants received pomalidomide 4 milligrams (mg) orally (PO) on Days 1 to 14 in each treatment cycle; bortezomib 1.3 mg/meter square (m^2) subcutaneous (SC) injection on Days 1, 4, 8 and 11 (Cycles 1 to 8) and on Days 1 and 8 (Cycle 9 onwards); and dexamethasone 20 mg (or 10 mg for participants aged greater than [>] 75 years) PO on Days 1, 2, 4, 5, 8, 9, 11 and 12 (Cycles 1 to 8) and Days 1, 2, 8 and 9 (Cycle 9 onwards). Each treatment cycle of 21 days. In daratumumab, pomalidomide and dexamethasone (DPd) treatment, participants received daratumumab 1800 mg SC injection weekly on Days 1, 8, 15 and 22 (Cycle 1 and 2), every 2 weeks on Days 1 and 15 (Cycle 3 to 6) and every 4 weeks on Day 1 (Cycle 7 onwards); pomalidomide 4 mg PO on Days 1 to 21 (Cycle 1 onwards); dexamethasone 40 mg (or 20 mg for participants aged >75 years) PO or intravenous(IV) weekly during Cycle 1-2 on Days 1, 8, 15, and 22 or split with 20 mg on Days 1, 2, 8, 9, 15, 16, 22, and 23. Each treatment cycle of 28 days. Participants continued to receive PVd or DPd until confirmed progressive disease (PD), death, intolerable toxicity, withdrawal of consent, or end of study, whichever occurred earlier.
- Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel]): Participants received at least one cycle of bridging therapy, that is PVd: pomalidomide 4 mg PO on Days 1 to 14, bortezomib 1.3 mg/m^2 SC injection on Days 1, 4, 8, and 11, and dexamethasone 20 mg (or 10 mg for participants aged >75 years) PO on Days 1, 2, 4, 5, 8, 9, 11, and 12; each treatment cycle of 21 days. DPd: daratumumab SC 1800 mg (co-formulated with rHuPH20) weekly on Days 1, 8, 15, and 22, pomalidomide 4 mg PO on Days 1 to 21, and dexamethasone PO or IV 40 mg (or 20 mg for participants aged >75 years) weekly during Cycle 1-2 on Days 1, 8, 15, and 22 or split with 20 mg on Days 1, 2, 8, 9, 15, 16, 22, and 23. Each treatment cycle of 28 days. Additional cycles of bridging therapy was considered based on participant's clinical status and timing of availability of JNJ-68284528 (cilta-cel). Followed by bridging therapy, participants received conditioning regimen: cyclophosphamide 300 mg/m^2 IV and fludarabine 30 mg/m^2 IV daily, for 3 days on chimeric antigen receptor T cells (CAR-T) Day -5, -4, -3 (prior to JNJ-68284528 infusion), followed by JNJ-68284528 (cilta-cel) infusion 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T cells per kilogram (kg) 5 to 7 days after the start of conditioning regimen.
Period: Overall Study
Arm/Group | Arm A: Standard Therapy: PVd or DPd | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel])
Started | 211 | 208
Treated (Safety Analysis Set) | 208 | 208
Completed | 0 | 0
Not Completed | 211 | 208
Not completed — Ongoing | 124 | 157
Not completed — Death | 82 | 50
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Standard Therapy: PVd or DPd | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel]) | Total
Number analyzed (Participants) | 211 | 208 | 419
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (9.09) | 59.7 (10.09) | 60.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 92 | 179
  Male | 124 | 116 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 165 | 152 | 317
  Unknown or Not Reported | 36 | 38 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 20 | 16 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 157 | 157 | 314
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: defined as time from date of randomization to date of first documented progressed disease (PD) as per International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurred first. PD: increase of 25% from lowest response value: serum and urine M-component (absolute increase must be >=0.5 grams per deciliter [g/dL] and >=200 milligrams [mg] per 24 hours, respectively); only in participants without measurable serum and urine M-protein levels, difference between involved and uninvolved free light chain (FLC) levels (absolute increase of >10 mg/dL); only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell (PC)% (absolute increase of >=10%), appearance of new lesion; definite development of new bone lesions or definite increase in size of existing bone lesions, >=50% increase in circulating PCs (minimum of 200 cells per microliter [uL]) if this was only measure of disease.
Time Frame: From randomization (Day 1) to either progressive disease or death, whichever occurred first (up to 3.9 years)
Population: The intent-to-treat (ITT) analysis set included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Standard Therapy: PVd or DPd | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel])
Number analyzed (Participants) | 211 | 208
months | 11.79 [9.66 to 14.00] | NA [34.50 to NA] — NA refers to data not estimable for median and upper limit of 95% confidence interval due to insufficient number of participants with events.

2. Secondary Outcome: Percentage of Participants Who Achieved Complete Response (CR) or Stringent Complete Response (sCR)
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

3. Secondary Outcome: Percentage of Participants Who Achieved Overall Minimal Residual Disease (MRD) Negative Status (at 10^-5)
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

4. Secondary Outcome: Percentage of Participants Who Were in CR or sCR and Achieved MRD-negative Status at 12 Months +/-3 Months
Time Frame: From randomization (Day 1) up to 12 months +/- 3 months
Reporting Status: Not Posted, anticipated posting 2028-06

5. Secondary Outcome: Percentage of Participants Who Achieved Sustained MRD-negative Status
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

6. Secondary Outcome: Overall Survival (OS)
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

7. Secondary Outcome: Time to Worsening of Symptoms Using the Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) Total Symptom Score
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

8. Secondary Outcome: Overall Response Rate (ORR)
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

9. Secondary Outcome: Progression Free Survival on Next-line Therapy (PFS2)
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Time Frame: From Cycle 1 Day 1 up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) by Severity
Time Frame: From Cycle 1 Day 1 up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

12. Secondary Outcome: Change From Baseline in Systemic Cytokine Concentrations on Participants Who Received Cilta-cel as Study Treatment (Arm B)
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

13. Secondary Outcome: Change From Baseline in Levels of CAR-T Cell Activation Markers on Participants Who Received Cilta-cel as Study Treatment (Arm B)
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

14. Secondary Outcome: Change From Baseline in Levels of JNJ-68284528 T Cell Expansion (Proliferation), and Persistence on Participants Who Received Cilta-cel as Study Treatment (Arm B)
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

15. Secondary Outcome: Number of Participants With Anti-JNJ-68284528 Antibodies on Participants Who Received Cilta-cel as Study Treatment (Arm B)
Time Frame: From Cycle 1 Day 1 up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

16. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 Item (EORTC-QLQ-C30) Scale Score
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

17. Secondary Outcome: Change From Baseline in Health-Related Quality of Life as Assessed by MySIm-Q Scale Sore
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

18. Secondary Outcome: Change From Baseline in Health-Related Quality of Life as Assessed by European Quality of Life - 5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire Scale Score
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

19. Secondary Outcome: Change From Baseline in Health-Related Quality of Life as Assessed by Patient Global Impression of Symptom Severity (PGIS) Scale Score
Time Frame: From baseline (Cycle 1 Day 1) up to 7 years (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2028-06

20. Secondary Outcome: Number of Participants in Health-Related Quality of Life as Assessed by The Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Item
Time Frame: From randomization (Day 1) up to 7 years
Reporting Status: Not Posted, anticipated posting 2028-06

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization (Day 1) up to 3.9 years; SAEs/Other AEs: Arm A: From Cycle 1 Day 1 up to 45 months; Arm B: From Cycle 1 Day 1 up to 8 months
Description: All-cause mortality was analyzed on all randomized participants. Serious and other AEs were analyzed in safety analysis set that included all participants who received any part of study treatment.
Arm/Group | Arm A: Standard Therapy: PVd or DPd | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel])
All-Cause Mortality (participants affected / at risk) | 83/211 | 50/208
Serious Adverse Events (participants affected / at risk) | 98/208 | 98/208
Other Adverse Events (participants affected / at risk) | 207/208 | 208/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Standard Therapy: PVd or DPd (N=208) | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel]) (N=208)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Cytopenia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 5
Hyperviscosity Syndrome (Blood and lymphatic system disorders) | 1 | 0
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 1
Atrial Flutter (Cardiac disorders) | 1 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 3
Pyrexia (General disorders) | 5 | 4
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 1 | 7
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Pericarditis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Covid-19 (Infections and infestations) | 7 | 6
Covid-19 Pneumonia (Infections and infestations) | 12 | 12
Cytomegalovirus Chorioretinitis (Infections and infestations) | 2 | 0
Cytomegalovirus Colitis (Infections and infestations) | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 1 | 2
Cytomegalovirus Infection Reactivation (Infections and infestations) | 1 | 0
Device Related Sepsis (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Enterocolitis Viral (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Gastroenteritis Bacterial (Infections and infestations) | 0 | 1
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 | 1
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Haemophilus Sepsis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Jc Virus Infection (Infections and infestations) | 1 | 0
Large Intestine Infection (Infections and infestations) | 0 | 1
Leishmaniasis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2
Metapneumovirus Infection (Infections and infestations) | 1 | 0
Metapneumovirus Pneumonia (Infections and infestations) | 0 | 3
Neutropenic Sepsis (Infections and infestations) | 1 | 1
Parainfluenzae Virus Infection (Infections and infestations) | 4 | 1
Parvovirus B19 Infection (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 14 | 8
Pneumonia Haemophilus (Infections and infestations) | 1 | 0
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pneumonia Legionella (Infections and infestations) | 2 | 0
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 | 1
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Pseudomonal (Infections and infestations) | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 | 1
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 1 | 1
Post Procedural Infection (Infections and infestations) | 1 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 1 | 0
Pseudomonal Sepsis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1
Rhinovirus Infection (Infections and infestations) | 3 | 0
Rotavirus Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Septic Shock (Infections and infestations) | 1 | 0
Sinusitis Bacterial (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 2
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 1
Viral Uveitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tracheal Obstruction (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Procalcitonin Increased (Investigations) | 1 | 0
Troponin I Increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 5
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epstein-Barr Virus Associated Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Myelodysplastic Syndrome with Multilineage Dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm of Appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral T-Cell Lymphoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Serous Cystadenocarcinoma Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial Paralysis (Nervous system disorders) | 1 | 9
Facial Paresis (Nervous system disorders) | 0 | 1
Iiird Nerve Paralysis (Nervous system disorders) | 0 | 1
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 2 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 1
Subdural Hygroma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Trigeminal Palsy (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Mental Disorder (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 3 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Standard Therapy: PVd or DPd (N=208) | Arm B: JNJ-68284528 (Ciltacabtagene Autoleucel [Cilta-cel]) (N=208)
Anaemia (Blood and lymphatic system disorders) | 57 | 110
Leukopenia (Blood and lymphatic system disorders) | 16 | 27
Lymphopenia (Blood and lymphatic system disorders) | 29 | 47
Neutropenia (Blood and lymphatic system disorders) | 178 | 187
Thrombocytopenia (Blood and lymphatic system disorders) | 67 | 113
Cataract (Eye disorders) | 15 | 1
Vision Blurred (Eye disorders) | 12 | 4
Abdominal Pain (Gastrointestinal disorders) | 16 | 10
Constipation (Gastrointestinal disorders) | 47 | 49
Diarrhoea (Gastrointestinal disorders) | 65 | 69
Nausea (Gastrointestinal disorders) | 43 | 101
Vomiting (Gastrointestinal disorders) | 18 | 29
Asthenia (General disorders) | 34 | 36
Chills (General disorders) | 8 | 13
Fatigue (General disorders) | 70 | 60
Oedema Peripheral (General disorders) | 28 | 35
Pyrexia (General disorders) | 31 | 31
Cytokine Release Syndrome (Immune system disorders) | 0 | 129
Hypogammaglobulinaemia (Immune system disorders) | 18 | 94
Bronchitis (Infections and infestations) | 21 | 4
Covid-19 (Infections and infestations) | 61 | 16
Nasopharyngitis (Infections and infestations) | 21 | 12
Pneumonia (Infections and infestations) | 12 | 8
Respiratory Tract Infection (Infections and infestations) | 17 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 51 | 21
Urinary Tract Infection (Infections and infestations) | 14 | 10
Fall (Injury, poisoning and procedural complications) | 12 | 9
Alanine Aminotransferase Increased (Investigations) | 15 | 17
Aspartate Aminotransferase Increased (Investigations) | 7 | 11
Blood Alkaline Phosphatase Increased (Investigations) | 4 | 11
Gamma-Glutamyltransferase Increased (Investigations) | 3 | 14
Decreased Appetite (Metabolism and nutrition disorders) | 13 | 34
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 39
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 32
Back Pain (Musculoskeletal and connective tissue disorders) | 46 | 31
Bone Pain (Musculoskeletal and connective tissue disorders) | 23 | 21
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 31 | 21
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 14 | 8
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 22 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 14
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 16 | 17
Dizziness (Nervous system disorders) | 30 | 24
Headache (Nervous system disorders) | 27 | 55
Paraesthesia (Nervous system disorders) | 10 | 12
Peripheral Sensory Neuropathy (Nervous system disorders) | 43 | 33
Tremor (Nervous system disorders) | 22 | 14
Anxiety (Psychiatric disorders) | 13 | 9
Insomnia (Psychiatric disorders) | 55 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 43 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 19
Rash (Skin and subcutaneous tissue disorders) | 11 | 22
Hypertension (Vascular disorders) | 21 | 15
Hypotension (Vascular disorders) | 2 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT04181827/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04181827/SAP_001.pdf